CLINICAL TRIAL: NCT05393973
Title: Effects of Core Stability Versus Swiss Ball Exercise Program on Pain, Range of Motion and Function in Patients With Chronic Neck Pain
Brief Title: Effects of Core Stability Versus Swiss Ball Exercise in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0145 Yumna
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Neck Pain
Keywords: Neck pain; Posture; Range of motion; Core Stability
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core stability exercises along with conventional physical therapy (Experimental): Core stability exercises
  Interventions: Other: Core stability exercises along with conventional physical therapy
- Swiss ball exercises along with the conventional physical therapy protocol (Experimental): Swiss ball exercises
  Interventions: Other: Swiss ball exercises along with the conventional physical therapy protocol

INTERVENTIONS:
Other: Core stability exercises along with conventional physical therapy — Core stability exercises included neck isometric exercises(flexion, extension, lateral flexion, rotation), chin tuck, chin tuck into towel, cervical extension + 10 minutes hot pack+ 10 minutes stretching (cervical flexors, extensors, rotators), session will be of 30-40 minutes, three times a week, for 4 weeks duration.
  Chin Tuck: In standing subject pulls back the chin( as if trying to make a double chin) while keeping the eyes level. This will be done for 15 repetitions.
  Cervical extension: In a standing position, the subject grasps the base of the neck, with both hands while extending the neck as far as possible. This will be done for 15 repetitions
  Arms: Core stability exercises along with conventional physical therapy
Other: Swiss ball exercises along with the conventional physical therapy protocol — Swiss ball exercise will be executed in the following order, assume supine posture on the treatment bed by fully extending their legs and putting them back on the bed in the most comfortable posture with hands on the abdomen. Second, while in the supine posture, support the head with one hand and insert a small Swiss ball near the back of the head with the other hand. Third, after having contacted the ball to the area below the back of the head, slowly turn the head and neck in the shape of the number '8'. Fourth, after having set 3 repetitions of rotating the head and neck for 10 seconds and then taking 10 seconds of general resting as 1 set of exercise, a total of 3 sets of exercise were executed with 1 minute of general resting taken between each set of exercise. Then perform neck flexion, extension, side bending, and rotation, hold each movement for 10 seconds + Hot pack (10 minutes) + 10 minutes of cervical stretching. Perform the exercise three times a week for 4 weeks duration.
  Arms: Swiss ball exercises along with the conventional physical therapy protocol

SUMMARY:
The study will be a randomized clinical trial to determine the effects of core stability versus swiss ball exercises on pain, range of motion and function in patients with chronic neck pain. A sample of 42 patients having neck pain since last 3 months will be taken from physical therapy department of "Bahawalpur medical & dental hospital" and will be divided into two groups each with 21 patients. Patient of any gender(male or female) with no history of neck surgery or any systemic disease will be considered. Group A will receive core stability exercises along with conventional physical therapy while group B will receive swiss ball exercises along with the conventional physical therapy protocol. The conventional physical therapy protocol will include a hot pack, and cervical stretches. The session will be around 30-45 minutes for each patient with three sessions per week on alternate days. A total of four-week treatment regime will be given to the patients and an assessment of patient's pain, range of motion, and function with NPRS (numeric pain rating scale), goniometry, and NDI (neck disability index) will be done at the baseline and after 4 weeks of treatment, data will be analyzed by using SPSS version 21, after the completion of treatment at four weeks.

DETAILED DESCRIPTION:
Chronic neck pain is one of the pains with the highest prevalence these days due to the imprecise daily life routine of people including students & office workers etc. It is generally declared that pain and stiffness in neck occur due to faulty posture for prolonged periods of time against the gravity. Deep layered muscles e.g longus capitus, longus Colli, rectus capitus anterior & rectus capitus lateralis provides the stability to neck if they are targeted it is believed that the observed problem can be cured. This study is aimed to compare two methods for stability of neck i.e. core stability exercises & swiss ball exercises.

Until now many treatment options have been used for chronic neck pain e.g stretching, isometrics, fascia release, mobilization techniques etc, and in recent literature, it is seen that stability of neck muscles are emerging to alleviate chronic neck pain. This study is aiming to compare the effects of core stability exercises and swiss ball exercises.So, the latest , effective and economical options for treatment can be used by the physical therapists and can be guided to the patients in order to gain long-lasting effects.

ELIGIBILITY:
Inclusion Criteria:

* • Both genders (male & female)

  * Age group 20-40 years
  * History of neck pain for more than 3 months

Exclusion Criteria:

* History of any neck surgery
* Neoplasms
* Any systemic disease
* Bony disorders

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
NPRS | 4th week
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain.
NDI | 4th week
  The NDI has become a standard instrument for measuring self-rated disability due to neck pain. Each of the 10 items scores from 0 to 5. The maximum score is 50
Goniometric measurement of neck ROM | 4th Week
  A goniometer is an instrument which measures the available range of motion at a joint.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil-ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- Bhawalpur Medical & Dental College, Bhawalpur, Chak Four Hundred Fifty-four, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta BD, Aggarwal S, Gupta B, Gupta M, Gupta N. Effect of Deep Cervical Flexor Training vs. Conventional Isometric Training on Forward Head Posture, Pain, Neck Disability Index In Dentists Suffering from Chronic Neck Pain. J Clin Diagn Res. 2013 Oct;7(10):2261-4. doi: 10.7860/JCDR/2013/6072.3487. Epub 2013 Oct 5. PMID 24298492
- [Background] Hoy DG, Protani M, De R, Buchbinder R. The epidemiology of neck pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):783-92. doi: 10.1016/j.berh.2011.01.019. PMID 21665126
- [Background] Kim BJ. Effects of Neck Stabilization and Swiss Ball Exercises on the Recovery from Fatigue of Neck Muscles in Turtle Neck Posture: Preliminary Experimental Study. Journal of International Academy of Physical Therapy Research. 2018;9(2):1498-507.
- [Background] Noormohammadpour P, Kordi M, Mansournia MA, Akbari-Fakhrabadi M, Kordi R. The Role of a Multi-Step Core Stability Exercise Program in the Treatment of Nurses with Chronic Low Back Pain: A Single-Blinded Randomized Controlled Trial. Asian Spine J. 2018 Jun;12(3):490-502. doi: 10.4184/asj.2018.12.3.490. Epub 2018 Jun 4. PMID 29879777
- [Background] Rajalaxmi V, Manickam M, Srilakshmi M, Arunselvi J, Jayabarathi R, Anupreethi P, et al. The role of multistep core stability exercise with and without conventional neck exercises in the treatment of chronic non-specific neck pain a randomized controlled trial. Biomedicine. 2020;40(2):232-5.
- [Background] He Y, Sun W, Zhao X, Ma M, Zheng Z, Xu L. Effects of core stability exercise for patients with neck pain: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2019 Nov;98(46):e17240. doi: 10.1097/MD.0000000000017240. PMID 31725601
- [Background] Ahn JA, Kim JH, Bendik AL, Shin JY. Effects of stabilization exercises with a Swiss ball on neck-shoulder pain and mobility of adults with prolonged exposure to VDTs. J Phys Ther Sci. 2015 Apr;27(4):981-4. doi: 10.1589/jpts.27.981. Epub 2015 Apr 30. PMID 25995537
- [Background] Cho H-Y, Park Y-J, Moon H-H, Park S-S, Kang G-M, Yoon W-Y, et al. The effect of swiss ball stabilisation exercise on deep and superficial cervical muscle and pain in patients with chronic neck pain. Indian Journal of Science and Technology. 2015;8:14.
- [Background] Correa EC, Berzin F. Mouth Breathing Syndrome: cervical muscles recruitment during nasal inspiration before and after respiratory and postural exercises on Swiss Ball. Int J Pediatr Otorhinolaryngol. 2008 Sep;72(9):1335-43. doi: 10.1016/j.ijporl.2008.05.012. Epub 2008 Jul 7. PMID 18603307